CLINICAL TRIAL: NCT03335761
Title: InterStim® Amplitude Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: MDT17030
Record Dates: First submitted 2017-10-23; First posted 2017-11-08 (Actual); Results first posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-12

CONDITIONS: Urinary Urge Incontinence
Keywords: Urinary; Incontinence
MeSH Terms: conditions — Urinary Incontinence, Urge

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Amplitude Setting #1 (Experimental): InterStim Therapy will be set to amplitude parameter #1.
  Interventions: Device: InterStim Therapy
- Amplitude Setting #2 (Experimental): InterStim Therapy will be set to amplitude parameter #2.
  Interventions: Device: InterStim Therapy
- Amplitude Setting #3 (Experimental): InterStim Therapy will be set to amplitude parameter #3.
  Interventions: Device: InterStim Therapy

INTERVENTIONS:
Device: InterStim Therapy — Device Programming

SUMMARY:
This feasibility study will explore the effects of three different InterStim amplitude settings on overactive bladder symptoms (OAB).

DETAILED DESCRIPTION:
This is a prospective, randomized, multicenter, single-blinded study to explore the efficacy and quality of life (QoL) of 3 different amplitude settings.

ELIGIBILITY:
Inclusion Criteria:

1. Primary diagnosis of urinary urge incontinence (UUI) as demonstrated on a 3-day baseline voiding diary demonstrating at least 3 UUI episodes
2. Female subjects 18 years of age or older
3. Candidate for InterStim Lead Placement
4. Willing and able to accurately complete voiding diaries, questionnaires, attend visits, and comply with the study protocol (which includes maintenance of InterStim II programming settings over the course of the study)
5. Willing and able to provide signed and dated informed consent
6. Willing to maintain current regimen (dosage and frequency) of any overactive bladder (OAB) medication

Exclusion Criteria:

1. Have neurological conditions such as multiple sclerosis, clinically significant peripheral neuropathy or spinal cord injury
2. History of diabetes unless the diabetes is well-controlled through diet and/or medications
3. Symptomatic urinary tract infection (UTI)
4. Have primary stress incontinence or mixed incontinence where the stress component overrides the urge component
5. Treatment of urinary symptoms with botulinum toxin in the past 9 months or any plan to have botulinum toxin treatment during the study
6. Implanted with a neurostimulator, pacemaker, or defibrillator
7. Have knowledge of planned MRIs, diathermy, microwave exposure, high output ultrasonic exposure, or radio frequency (RF) energy exposure not included within the scanning conditions provided with the MRI Guidelines for InterStim Therapy
8. Women who are pregnant or planning to become pregnant
9. Characteristics indicating a poor understanding of the study or characteristics that indicate the subject may have poor compliance with the study protocol requirements.
10. Currently enrolled or planning to enroll in a potentially confounding clinical study during the course of the study (co-enrollment in concurrent studies is only allowed when documented pre-approval is obtained from the Medtronic study manager (or designee).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 97 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2019-11-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (12):
  - Academic Urology & Urogynecology of Arizona, Phoenix, Arizona
  - East Coast Institute for Research, Jacksonville, Florida
  - Pinellas Urology, St. Petersburg, Florida
  - Florida Urology Partners, Tampa, Florida
  - Minnesota Urology Fridley, Fridley, Minnesota
  - Minnesota Urology Woodbury, Woodbury, Minnesota
  - Adult Pediatric Urology and Urogynecology, Omaha, Nebraska
  - Urologic Research & Consulting, Englewood, New Jersey
  - Carolina Urology Partners, Concord, North Carolina
  - Chattanooga Hamilton County Hospital Authority d/b/a Erlanger Health System, Chattanooga, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Aurora Research Institute - Aurora West Allis Women's Pavilion, West Allis, Wisconsin
- UZ Leuven - Campus Gasthuisberg - Department Urology, Leuven, Belgium
- University Urology Associates, Toronto Western Hospital, Toronto, Ontario, Canada
- CHU Hôpitaux de Rouen - Hôpital Charles Nicolle, Rouen, France
- Azienda Ospedaliera Universitaria Integrata Verona, Verona, Italy
- Erasmus MC, Rotterdam, Netherlands
- University College London Hospitals NHS Foundation Trust - University College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 97 subjects enrolled in the study, 48 were randomized, 46 were implanted with a neurostimulator device, and 43 completed their 12 week follow-up visit before exiting the study. Nineteen were randomized to 50% of sensory threshold, 14 were randomized to 80% of sensory threshold, and 15 were randomized to sensory threshold.
Groups:
- Amplitude Setting #1 = 50% Sensory Threshold: InterStim Therapy will be set to amplitude parameter #1 (50% Sensory Threshold)
  InterStim Therapy: Device Programming
- Amplitude Setting #2 = 80% Sensory Threshold: InterStim Therapy will be set to amplitude parameter #2 (80% Sensory Threshold)
  InterStim Therapy: Device Programming
- Amplitude Setting #3 = Sensory Threshold: InterStim Therapy will be set to amplitude parameter #3 (Sensory Threshold)
  InterStim Therapy: Device Programming
Period: Overall Study
Arm/Group | Amplitude Setting #1 = 50% Sensory Threshold | Amplitude Setting #2 = 80% Sensory Threshold | Amplitude Setting #3 = Sensory Threshold
Started | 19 | 14 | 15
Implanted With a Neurostimulator Device | 18 | 14 | 14
Completed | 17 | 13 | 13
Not Completed | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Population: This summarizes demographics for subjects in the Randomized Subject Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Amplitude Setting #1 = 50% Sensory Threshold | Amplitude Setting #2 = 80% Sensory Threshold | Amplitude Setting #3 = Sensory Threshold | Total
Number analyzed (Participants) | 19 | 14 | 15 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (16) | 57.9 (16.1) | 56.7 (14.9) | 60 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 14 | 15 | 48
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.0 (5.7) | 36.3 (11.2) | 33.1 (6.4) | 32.8 (8.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Urinary Urge Incontinence (UUI) Episodes Per Day From Baseline to 12 Weeks.
Description: Symptoms related to OAB were evaluated using paper voiding diaries. Subjects were trained to complete the urinary voiding diaries for 3-days.
Time Frame: 12 weeks
Population: Complete Case Subject Set
Measure: Mean (Standard Deviation); unit: UUI episodes/day
Arm/Group | Amplitude Setting #1 = 50% Sensory Threshold | Amplitude Setting #2 = 80% Sensory Threshold | Amplitude Setting #3 = Sensory Threshold
Number analyzed (Participants) | 17 | 13 | 13
UUI episodes/day
  UUI episodes per day at Baseline | 4.4 (2.9) | 5.3 (3.1) | 5.1 (4.7)
  UUI episodes per day at 12 weeks | 1.4 (2.6) | 2.4 (3.0) | 1.5 (2.3)
  Change in UUI episodes per day from baseline to 12 weeks | -3 (2.6) | -2.9 (2.9) | -3.6 (2.8)

2. Secondary Outcome: Change in QoL Using ICIQ-OAB QOL From Baseline to 12 Weeks.
Description: International Consultation on Incontinence Modular Questionnaire - Overactive Bladder Symptoms Quality of Life Questionnaire The questionnaire consists of 4 subscales and a single item on urinary symptom interference.
  The four subscales of Concern (7 items), Coping (8 items), Sleep (5 items), and Social (5 items) are measured on a scale from 0-100 using a range percentile transformation on the summed value from individual listed items. The Health-Related Quality of Life (HRQL) score is a calculated score with a range from 0 to 100 using a range percentile transformation on the summed value from the subscales. Subjects were asked a urinary symptom interference question. "Interference" was measured on a scale from 0-10.
  A positive change in Concern, Coping, Sleep, Social, and HRQL indicates improvement in Quality of Life; a negative change in Interference indicates improvement in Quality of Life.
Time Frame: 12 weeks
Population: Complete Case Subject Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Amplitude Setting #1 = 50% Sensory Threshold | Amplitude Setting #2 = 80% Sensory Threshold | Amplitude Setting #3 = Sensory Threshold
Number analyzed (Participants) | 17 | 13 | 13
units on a scale
  Change in Coping from baseline to 12 weeks | 44.4 (30.4) | 41.0 (26.3) | 39.4 (27.9)
  Change in Concern from baseline to 12 weeks | 48.2 (28.9) | 50.3 (17) | 49.9 (30.2)
  Change in Sleep from baseline to 12 weeks | 31.4 (26.6) | 37.8 (22.7) | 32.0 (31.6)
  Change in Social from baseline to 12 weeks | 20.9 (25.0) | 28.6 (17) | 20.6 (19.9)
  Change in HRQL from baseline to 12 weeks | 38.1 (24.4) | 40.5 (16.7) | 37.1 (23.4)
  Change in Interference from baseline to 12 weeks | -5.2 (3.3) | -4.7 (3.0) | -4.7 (3.5)

ADVERSE EVENTS:
Time Frame: From Post-Neurostimulator device implant to 12 weeks follow-up visit
Description: Serious, device related, procedure related, and/or therapy related adverse events are considered reportable for this study
Arm/Group | Amplitude Setting #1 = 50% Sensory Threshold | Amplitude Setting #2 = 80% Sensory Threshold | Amplitude Setting #3 = Sensory Threshold
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 3/19 | 1/14 | 3/15
Other Adverse Events (participants affected / at risk) | 3/19 | 1/14 | 3/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amplitude Setting #1 = 50% Sensory Threshold (N=19) | Amplitude Setting #2 = 80% Sensory Threshold (N=14) | Amplitude Setting #3 = Sensory Threshold (N=15)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amplitude Setting #1 = 50% Sensory Threshold (N=19) | Amplitude Setting #2 = 80% Sensory Threshold (N=14) | Amplitude Setting #3 = Sensory Threshold (N=15)
Medical device site pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/61/NCT03335761/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/61/NCT03335761/SAP_001.pdf